CLINICAL TRIAL: NCT07131800
Title: Objective and Perceptual Characteristics of the Voice After Endotracheal Intubation in Head and Neck Surgery
Acronym: VOICE
Status: Enrolling by invitation | Type: Observational
Sponsor: Clinical Hospital Centre Zagreb (Other)
Responsible Party: Principal Investigator, Renata Curić Radivojević, Primarius; MD; PhD; FESAIC, Clinical Hospital Centre Zagreb
Other Study IDs: Klasa8.1-23/209-3;Broj02/013AG
Record Dates: First submitted 2025-07-08; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Voice Disorder Due to Iatrogenic Factor; Endotracheal Intubation During Surgery; Thyroid Surgery; Head and Neck Surgery
Keywords: endotracheal intubation; surgery; head and neck; voice disorder; VHI
MeSH Terms: conditions — Voice Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients undergoing thyroid surgery: Patients undergoing scheduled thyroid surgery at the University Hospital Centre Zagreb under general endotracheal anesthesia without preoperative voice disorder regardless of the cause (previous operations or irradiation on the neck, and damage to the recurrent laryngeal nerve (RLN) during thyroidectomy).
- Patients undergoing abdominal surgery: Patients undergoing scheduled abdominal surgery at Day surgery of University Hospital Centre Zagreb under general anesthesia without preoperative voice disorder regardless of the cause (previous operations or irradiation on the neck, and damage to the recurrent laryngeal nerve (RLN) during thyroidectomy). This will include laparoscopic abdominal procedures and other minor abdominal procedures done in Day surgery, and will be control group for head and neck surgical procedures.
- Patients undergoing other head and neck surgery besides thyroid: Patients undergoing scheduled head and neck surgeries beside thyroid surgery at the University Hospital Centre Zagreb under general endotracheal anesthesia without preoperative voice disorder regardless of the cause (previous operations or irradiation on the neck, and damage to the recurrent laryngeal nerve (RLN) during thyroidectomy).

SUMMARY:
Introduction: Possible consequences of endotracheal intubation are post-intubation voice changes.

Hypothesis: Endotracheal intubation during head and neck surgery is associated with objective and perceptual voice disorders.

Research objective: To investigate the short-term and long-term effects of endotracheal intubation on voice quality during head and neck surgery.

Material, subjects, methodology and research design: A prospective observational cohort study that will include patients undergoing surgery and endotracheal intubation lasting up to 3 hours. Adult patients divided into three groups will be included in the research: thyroid surgery, parotid gland surgery and abdominal surgery. Videostroboscopy, perceptual and objective acoustic voice analysis will be recorded before surgery, on the second postoperative day, two weeks and 1 month after surgery.

Expected scientific contribution of the proposed research: The scientific contribution would be an understanding of the risk factors and the connection of voice disorders after endotracheal intubation, as well as the ability to determine differences in this risk in patients undergoing different operations.

DETAILED DESCRIPTION:
study protocol has been published and is attached below

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for elective thyroid, head and neck surgery or abdominal surgery
* 18 and 70 years,
* normal preoperative voice status, and
* normal laryngeal status.

Exclusion Criteria:

* <18 years in the time of surgery
* history of previous head and neck operation or radiotherapy
* patients scheduled for head and neck operation that can alter acoustic characteristics of the voice (surgery of the nasal cavity, ear surgery, laryngeal surgery, jaw surgery).
* Patients with preoperatively diagnosed pathologic vocal cord findings (nodules, polyps, vocal cord paralysis),
* patients with postoperative injuries of the vocal cords, recurrent and superior laryngeal nerve,
* patients with laryngopharyngeal reflux,
* patients in whom postoperative evaluation of the voice cannot be performed due to uncooperativeness will also be excluded from the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective thyroid, head and neck surgery or abdominal surgery at the University Hospital Centre Zagreb. All eligible patients will be divided into three groups, as follows: patients scheduled for thyroid gland surgery; patients scheduled for some other type of head and neck operation that does not fall to exclusion criteria (parotidectomy, extirpation of congenital neck cyst, etc.); and control group including patients scheduled for operation other than the head and neck region. All operations will be performed by experienced operators with more than 100 annual procedures.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-09-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Subjective analysis of voice changes before and after endotracheal intubation for thyroid surgery, other head and neck surgery and abdominal surgery using Voice Handicap Index (VHI) | Preoperative (within 7 days before surgery), Postoperative Day 1, Week 2, and Week 4
  The Voice Handicap Index (VHI) is one of the most frequently used self-assessment scales for voice disorders. The Croatian version was adapted and validated by Bonetti and Bonetti (2013), while Benšić et al. (2024) confirmed normative values for the Croatian language. The scale consists of 30 items divided into three subscales:
  - Functional, emotional and physical component. Each item is rated on a 5-point Likert scale (0 = Never, 1 = Almost Never, 2 = Sometimes, 3 = Almost Always, 4 = Always), giving a total score from 0 to 120, with higher scores indicating greater perceived voice handicap. Participants will complete the VHI questionnaire at Baseline (within 7 days before surgery with endotracheal intubation) and at postoperative follow-up time points (Day 1, Week 2, and Week 4).
  The primary VHI outcome is the change in total score before and after surgery.
  Units of Measure:
  • Total score range: 0-120
  Method of Administration:
  • Self-administered paper
Subjective analysis of voice changes before and after endotracheal intubation for thyroid surgery, other head and neck surgery and abdominal surgery using GRBAS Scale (Perceptual Voice Evaluation) | Time Points: Preoperative (within 7 days before surgery), Postoperative Day 1, Week 2, and Week 4
  The perceptual voice assessment (GRBAS) will be conducted by two speech-language pathologists with several years of clinical experience. Each parameter-Grade, Roughness, Breathiness, Asthenia, and Strain-will be scored on a 4-point scale (0 = Normal, 1 = Slight, 2 = Moderate, 3 = Severe). The average of the two evaluators' scores will be taken, and in the case of significant discrepancies, a third evaluator will be consulted to reach consensus.
  Voice samples will be recorded at baseline and post-intervention at 4 time points total. The primary GRBAS outcome will be the change in the 'Grade' score; secondary analyses will include changes in R, B, A, and S.
  Units of Measure:
  • Ordinal scores (0-3) for each parameter
Videostroboscopy Evaluation before and after surgery | Preoperative (within 7 days before surgery) and Postoperative day 1
  Videostroboscopy uses an endoscope containing a built-in video camera and a stroboscope, which records phonation while the vocal cords are being filmed. The recording captures the frequency of vocal cord vibrations during voice production and provides an apparently slow-motion view of these vibrations. In the stroboscopic video, the movements of the vocal cords are slowed down enough to precisely follow their motion. This technique allows detailed observation of the amplitude and symmetry of vibrations, as well as the phase of vocal cord closure during voice production. It facilitates diagnosis of numerous physical problems with the vocal cords, including paresis resulting from injury to the recurrent laryngeal nerve. Evaluations will be performed pre- and post-intervention using a standardized protocol. 2 experienced phoniatrists will independently review the recordings to identify possible pathology in vocal fold motion or structural damage. No formal scoring system will be applied.
Objective Acoustic and Aerodynamic Voice Analysis - changes in fundamental frequency before and after surgery | Time Points: Preoperative (within 7 days before surgery), Postoperative Day 1, Week 2, and Week 4
  Objective voice evaluation will be performed using selected acoustic and aerodynamic measures. Voice assessment involves recording sustained phonation of the vowel /a/ in a sound-treated room using a calibrated digital recording system. The recordings will be acquired with a high-quality microphone positioned at a fixed distance of 30 cm from the participant's mouth, placed at a 45° angle. The sound signal will be analyzed using the LingWAVES SLP Suite Pro VPR software (WEVOSYS medical technology GmbH, Germany). This software converts the analog voice signal to digital form and processes it to extract relevant voice parameters.
  Parameters to be evaluated:
  • Fundamental frequency (F0) in Hz.
  Physiological reference values:
  • Fundamental frequency: Female: ~206 Hz, Male: ~120 Hz,

SECONDARY OUTCOMES:
Objective Acoustic and Aerodynamic Voice Analysis - changes in Intensity before and after surgery | Time Points: Preoperative (within 7 days before surgery), Postoperative Day 1, Week 2, and Week 4
  Objective voice evaluation will be performed using selected acoustic and aerodynamic measures. Voice assessment involves recording sustained phonation of the vowel /a/ in a sound-treated room using a calibrated digital recording system. The recordings will be acquired with a high-quality microphone positioned at a fixed distance of 30 cm from the participant's mouth, placed at a 45° angle.
  The sound signal will be analyzed using the LingWAVES SLP Suite Pro VPR software (WEVOSYS medical technology GmbH, Germany). This software converts the analog voice signal to digital form and processes it to extract relevant voice parameters.
  Parameters to be evaluated:
  • Intensity (in dB)
  Physiological reference values:
  • Intensity: Female: 68-74 dB, Male: 68-76 dB
Objective Acoustic and Aerodynamic Voice Analysis- changes in Jitter before and after surgery | Time Points: Preoperative (within 7 days before surgery), Postoperative Day 1, Week 2, and Week 4
  Objective voice evaluation will be performed using selected acoustic and aerodynamic measures. Voice assessment involves recording sustained phonation of the vowel /a/ in a sound-treated room using a calibrated digital recording system. The recordings will be acquired with a high-quality microphone positioned at a fixed distance of 30 cm from the participant's mouth, placed at a 45° angle.
  The sound signal will be analyzed using the LingWAVES SLP Suite Pro VPR software (WEVOSYS medical technology GmbH, Germany). This software converts the analog voice signal to digital form and processes it to extract relevant voice parameters.
  Parameters to be evaluated:
  • Jitter (%)
  Physiological reference values:
  • Jitter: 0-0.5%
Objective Acoustic and Aerodynamic Voice Analysis- changes in shimmer before and after surgery | Time Points: Preoperative (within 7 days before surgery), Postoperative Day 1, Week 2, and Week 4
  Objective voice evaluation will be performed using selected acoustic and aerodynamic measures. Voice assessment involves recording sustained phonation of the vowel /a/ in a sound-treated room using a calibrated digital recording system. The recordings will be acquired with a high-quality microphone positioned at a fixed distance of 30 cm from the participant's mouth, placed at a 45° angle.
  The sound signal will be analyzed using the LingWAVES SLP Suite Pro VPR software (WEVOSYS medical technology GmbH, Germany). This software converts the analog voice signal to digital form and processes it to extract relevant voice parameters.
  Parameters to be evaluated:
  • Shimmer (%)
  Physiological reference values:
  • Shimmer: 0-5%
Objective Acoustic and Aerodynamic Voice Analysis- changes in Maximum phonation time before and after surgery | Time Points: Preoperative (within 7 days before surgery), Postoperative Day 1, Week 2, and Week 4
  Objective voice evaluation will be performed using selected acoustic and aerodynamic measures. Voice assessment involves recording sustained phonation of the vowel /a/ in a sound-treated room using a calibrated digital recording system. The recordings will be acquired with a high-quality microphone positioned at a fixed distance of 30 cm from the participant's mouth, placed at a 45° angle.
  The sound signal will be analyzed using the LingWAVES SLP Suite Pro VPR software (WEVOSYS medical technology GmbH, Germany). This software converts the analog voice signal to digital form and processes it to extract relevant voice parameters.
  Parameters to be evaluated:
  • Maximum phonation time (MPT, in seconds)
  Physiological reference values:
  • Maximum phonation time: Female: 15-25 sec, Male: 25-35 sec

CONTACTS AND LOCATIONS:
Overall Officials: Ivana Šimić Prgomet, PhD, mag.logoped, Professor log., Principal Investigator — Clinical Hospital Centre Zagreb; Drago Prgomet, MD; PhD, Professor, Study Director — Clinical Hospital Centre Zagreb; Renata Curić Radiovjević, Primarius, Study Chair — Clinical Hospital Centre Zagreb
Locations (1):
- University Hospital Centre Zagreb, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No
At the moment, we do not know other logopedic laboratory being able to perform the same audiometric evaluation.

REFERENCES:
- [Background] Simic I, Curic Radivojevic R, Slipac J, Prgomet D. VOICE CONDITION FOLLOWING SHORT-TERM ENDOTRACHEAL INTUBATION IN HEAD AND NECK SURGERY: STUDY PROTOCOL FOR CLINICAL TRIAL. Acta Clin Croat. 2023 Apr;62(Suppl1):49-54. doi: 10.20471/acc.2023.62.s1.06. PMID 38746618